CLINICAL TRIAL: NCT03934307
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Single Dose and Active Comparator-Controlled Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered ALN-AGT01 in Patients With Hypertension
Brief Title: A Study to Evaluate ALN-AGT01 in Patients With Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-AGT01-001; 2019-000129-39 (EudraCT Number)
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A: SAD: ALN-AGT01 (Experimental): Participants will be administered a single dose of ALN-AGT01.
  Interventions: Drug: ALN-AGT01
- Part A: SAD: ALN-AGT01-Matching Placebo (Placebo Comparator): Participants will be administered a single dose of ALN-AGT01-matching placebo.
  Interventions: Drug: ALN-AGT01-Matching Placebo
- Part B: SD: ALN-AGT01 (Experimental): Participants with controlled salt intake will be administered a single dose of ALN-AGT01.
  Interventions: Drug: ALN-AGT01
- Part B: SD: ALN-AGT01-Matching Placebo (Placebo Comparator): Participants with controlled salt intake will be administered a single dose of ALN-AGT01-matching placebo.
  Interventions: Drug: ALN-AGT01-Matching Placebo
- Part D: MD: ALN-AGT01 + Irbesartan-Matching Placebo (Experimental): Participants, who are obese, will be administered multiple doses of ALN-AGT01 and irbesartan-matching placebo.
  Interventions: Drug: ALN-AGT01; Drug: Irbesartan-Matching Placebo
- Part D: MD: ALN-AGT01-Matching Placebo + Irbesartan (Active Comparator): Participants, who are obese, will be administered multiple doses of ALN-AGT01-matching placebo and irbesartan.
  Interventions: Drug: ALN-AGT01-Matching Placebo; Drug: Irbesartan
- Part E: Open Label: ALN-AGT01 + Irbesartan (Experimental): Participants will be administered a single dose of ALN-AGT01 and multiple doses of irbesartan.
  Interventions: Drug: ALN-AGT01; Drug: Irbesartan

INTERVENTIONS:
Drug: ALN-AGT01 — ALN-AGT01 will be administered by subcutaneous (SC) injection.
  Other Names: Zilebesiran
  Arms: Part A: SAD: ALN-AGT01; Part B: SD: ALN-AGT01; Part D: MD: ALN-AGT01 + Irbesartan-Matching Placebo; Part E: Open Label: ALN-AGT01 + Irbesartan
Drug: ALN-AGT01-Matching Placebo — Normal saline (0.9% NaCl) matching volume of ALN-AGT01 doses will be administered SC.
  Arms: Part A: SAD: ALN-AGT01-Matching Placebo; Part B: SD: ALN-AGT01-Matching Placebo; Part D: MD: ALN-AGT01-Matching Placebo + Irbesartan
Drug: Irbesartan — Irbesartan will be administered orally.
  Arms: Part D: MD: ALN-AGT01-Matching Placebo + Irbesartan; Part E: Open Label: ALN-AGT01 + Irbesartan
Drug: Irbesartan-Matching Placebo — Irbesartan-matching placebo will be administered orally.
  Arms: Part D: MD: ALN-AGT01 + Irbesartan-Matching Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) effects of subcutaneous (SC) ALN-AGT01 (zilebesiran) in participants with hypertension. The study will be conducted in 4 parts: Part A will be a single ascending dose (SAD) phase in hypertensive participants, Part B will be a single dose (SD) phase in hypertensive participants with controlled salt intake, Part D will be a MD phase in hypertensive participants who are obese, and Part E will be an open-label SD phase with co-administration of irbesartan in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Has mild to moderate hypertension with mean sitting systolic blood pressure (SBP) of >130 and ≤165 mmHg without hypertensive medication for Parts A, B and D, and >135 and ≤165 mmHg without hypertensive medication for Part E
* Parts A and B: Has body mass index (BMI) ≥18 and ≤35 kg/m^2; Part D: Has BMI >35 and ≤50 kg/m^2; Part E: Has BMI ≥18 kg/m^2 and ≤50 kg/m^2
* Has a normal 12-lead electrocardiogram (ECG)
* Is a nonsmoker

Exclusion Criteria:

* Has secondary hypertension
* Has orthostatic hypotension
* Has estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73m^2
* Recently received an investigational agent
* Has diabetes mellitus
* Has history of any cardiovascular event
* Has history of intolerance to SC injection(s)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Parts A, B and E: each up to approximately 12 months; Part D: up to approximately 18 months

SECONDARY OUTCOMES:
Change from Baseline in Blood Angiotensinogen (AGT) Level | Parts A, B and E: each up to approximately 12 months; Part D: up to approximately 18 months
Maximum Observed Plasma Concentration (Cmax) of ALN-AGT01 and of Potential Metabolites | Parts A, B and E: Up to Day 15; Part D: Up to Day 99
Area Under the Concentration-time Curve (AUC) of ALN-AGT01 and of Potential Metabolites | Parts A, B and E: Up to Day 15; Part D: Up to Day 99

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (3):
- United Kingdom (3):
  - Clinical Trial Site, Edinburgh
  - Clinical Trial Site, London
  - Clinical Trial Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badri P, Kolachana K, Duong A, Lasko M, Nandi T, Mehrotra N, Robbie GJ. Platform Assessment of Concentration-QTc Relationship Across GalNAc-siRNA Molecules. Clin Pharmacokinet. 2025 Dec 12. doi: 10.1007/s40262-025-01606-0. Online ahead of print. PMID 41388232
- [Derived] Desai AS, Webb DJ, Taubel J, Casey S, Cheng Y, Robbie GJ, Foster D, Huang SA, Rhyee S, Sweetser MT, Bakris GL. Zilebesiran, an RNA Interference Therapeutic Agent for Hypertension. N Engl J Med. 2023 Jul 20;389(3):228-238. doi: 10.1056/NEJMoa2208391. PMID 37467498